CLINICAL TRIAL: NCT02928068
Title: Telehealth Coaching for Families of Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00002264
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Autism Spectrum Disorders
Keywords: telehealth
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Occupational Performance Coaching (OPC) (Experimental): This group received approximately 12 sessions of the telehealth intervention. The intervention consisted of parent-therapist conversations via telehealth to increase child function and participation.
  Interventions: Behavioral: Occupational Performance Coaching (OPC)

INTERVENTIONS:
Behavioral: Occupational Performance Coaching (OPC) — OPC focuses on increasing positive child-caregiver interactions and child learning opportunities in everyday routines and contexts, which positions families for improved trajectories over time. OPC capitalizes on families' strengths, while supporting caregivers in using their own resources and ideas to advance child function. Caregivers identify goals, while therapists ask reflective questions and make reflective comments, affording caregivers an opportunity to gain a deeper understanding of their own current knowledge and the impact of their strategies on their children's adaptive behavior. Thus, families generate their own solutions and are ultimately responsible for carrying out the intervention and evaluating its effectiveness.

SUMMARY:
The purpose of this study is to investigate the efficacy of a 12 week telehealth intervention for families of children with autism spectrum disorders under the age of 6 years on child participation and parent efficacy.

DETAILED DESCRIPTION:
Autism spectrum disorders (ASD) are increasingly being diagnosed in children, creating a pressing need for effective and cost-efficient models of early intervention (EI) services. Many EI systems are struggling to meet the needs of the increasing number of families of children with ASD. In rural areas, there is a shortage of EI therapists, and the distances to reach families results in an inefficient use of professional time and research shows that rural families of children with ASD receive fewer EI services, which has detrimental effects on children's developmental trajectories. If occupational therapy interventions for young children with ASD utilize innovative methods of service delivery in rural areas, investigators can increase the number of families that receive services thereby positively influencing child and family outcomes. Therefore, investigators propose to test the acceptability, cost-effectiveness, and efficacy of a 12 week telehealth intervention for families of young children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Family with a child up to 72 months old with a diagnosis of ASD and primarily spoke English in the home.

Exclusion Criteria:

* Child has significant visual or hearing impairments or has a known genetic condition associated with autism (e.g., Fragile X Syndrome).

Ages: 12 Months to 84 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2015-04; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Parent Sense of Competence Scale | 12 weeks

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Little, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- Occupational Therapy Education, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Little LM, Pope E, Wallisch A, Dunn W. Occupation-Based Coaching by Means of Telehealth for Families of Young Children With Autism Spectrum Disorder. Am J Occup Ther. 2018 Mar/Apr;72(2):7202205020p1-7202205020p7. doi: 10.5014/ajot.2018.024786. PMID 29426380